CLINICAL TRIAL: NCT06217237
Title: Phase II Neuroimaging Network: Optimization and Harmonization of Advanced MRI Sequences and Their Application in the Study of Dementia and Intellectual Disability in Pediatric Age
Brief Title: Optimization and Harmonization of Advanced MRI Sequences
Status: Completed | Type: Observational
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Sponsor
Other Study IDs: RETEimaging_IRCCS_001
Record Dates: First submitted 2023-03-21; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2023-10

CONDITIONS: Dementia Frontal; Dementia Alzheimers; Lewy Body Variant of Alzheimer Disease; Neuro-Degenerative Disease
MeSH Terms: conditions — Alzheimer Disease; Lewy Body Variant of Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AD FDT DBL GROUP: All participants will undergo an MRI session. The MRI protocol will include the clinical diagnostic protocol defined within the Network and research sequences as specified above (T1 3D, DTI, FLAIR 3D, QSM).
  Interventions: Diagnostic Test: AD FDT DBL GROUP
- CONTROL GROUP: All participants will undergo an MRI session. The MRI protocol will include the clinical diagnostic protocol defined within the Network and research sequences as specified above (T1 3D, DTI, FLAIR 3D, QSM).

INTERVENTIONS:
Diagnostic Test: AD FDT DBL GROUP — All participants will undergo an MRI session. The MRI protocol will include the clinical diagnostic protocol defined within the Network and research sequences as specified above (T1 3D, DTI, FLAIR 3D, QSM).
  Groups: AD FDT DBL GROUP

SUMMARY:
Development of a shared multimodal MRI protocol for the definition and quantification of imaging biomarkers in AD, DLB, FDT dementias, especially white matter alterations.

DETAILED DESCRIPTION:
Development of a shared multimodal MRI protocol for the definition and quantification of imaging biomarkers in AD, DLB, FDT dementias, especially white matter alterations.

ELIGIBILITY:
Inclusion Criteria:

for patients

* accident cases
* time of onset of NOT MORE THAN 24 months
* Clinical Dementia Rating Scale (CDR) <=2;
* MoCA<=17

for controls absence of complaints of cognitive disorders and/or neurological/neuropsychological visits for the evaluation of such disorders;

* CDR = 0;
* MoCA>=27. for all Age >= 50 and <= 80;
* Hachinski Ischemic Scale - 7 items < 2;
* visual and/or auditory acuity sufficient to carry out the neuropsychological assessment;
* if on neuropsychopharmacological therapy, stability for 4 weeks before the start of the study.

Exclusion Criteria:

for all

* any uncontrolled medical condition or neurological/neurodegenerative disease that, in the opinion of the recruiting physician, could contribute to the individual's cognitive impairment [e.g., kidney disease, liver disease, brain tumor, alcohol or drug abuse, abnormal thyroid function, hydrocephalus normotensive, vascular dementia, neurocognitive disorder due to head trauma (according to the diagnostic criteria of the DSM V)];
* transient ischemic attack or stroke during the 12 months preceding screening; history of unstable angina, myocardial infarction, heart failure (New York Heart Association Class III or IV), or clinically significant heart rhythm disturbances documented within one year of screening;
* history of malignant tumor disease, except: cancer in remission for more than 5 years since screening; prostate cancer in situ;
* history of surgically treated squamous cell carcinoma or basal cell carcinoma;
* impaired liver function or liver failure;
* history or evidence of autoimmune disease considered clinically significant by the doctor or requiring the chronic use of corticosteroids or other immunosuppressive drugs;
* clinically significant systemic illness or infection within 30 days of screening; comorbidity for primary psychiatric or neurological disorders;
* absence of an informant (partner, relative, adult child or friend) who knows the subject well enough to be able to provide reliable information on his cognitive and functional abilities.
* contraindication to carrying out the MRI exam.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients and controls recruited based on the inclusion criteria carry out clinical and neuropsychological tests
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2021-01-10 (Actual)

PRIMARY OUTCOMES:
Quantitative Susceptibility Mapping (QSM), Diffusion Weighted Imaging (DWI) - Diffusion Tensor Imaging (DTI), Fluid Attenuated Inversion Recovery (FLAIR) | during MRI procedure
  The main endpoint is the characterization of white matter alterations in different forms of dementing diseases through the combined study of MRI sequences. Specifically, we correlate Voxel Based Morphometry indices, DTI quantifcation and lesions volume with MMSE and MOCA scores.

SECONDARY OUTCOMES:
FLAIR, QSM, DWI (DTI) for white matter study | during MRI procedureRMN date examination
  Quantitative analysis of FLAIR, QSM, DWI (DTI) for white matter evaluation
  ES2. Characterization of white matter alterations which will also take place through the quantification of:
  * microstructure and macrostructure values of the white matter through diffusion techniques (including DTI)
  * white matter lesions through post-processing algorithms (14) applied to the FLAIR sequence;
  * magnetic susceptibility in the white matter and in particular in myelin (15), through the QSM technique;
  ES3. Definition of an automatic single-case multimodal algorithm (MUQUBIA) for the quantification and classification of subjects with alterations of the white matter (as emerged from MRI data) useful for doctors in the Network.
  ES4. Evaluation of variables of interest emerging from MRI analyzes in relation to clinical and neuropsychological variables

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Centro Neurolesi "Bonino-Pulejo", Messina, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Corresponding author